CLINICAL TRIAL: NCT01882114
Title: Study of Atherosclerotic Risk Factors and Oxidative Stress in Atrial Fibrillation. Relation to Cardiovascular Events
Brief Title: Atherosclerosis in Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Pasquale Pignatelli, Associate Professor, University of Roma La Sapienza
Other Study IDs: MetS1306/2007
Record Dates: First submitted 2013-05-24; First posted 2013-06-20 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Atrial Fibrillation; Metabolic Syndrome; Oxidative Stress; Atherosclerosis; Disorders, Blood Coagulation
Keywords: atherosclerosis; cardiovascular events; ankle-brachial index; carotid disease; echocardiography; mediterranean diet; platelet activation
MeSH Terms: conditions — Atrial Fibrillation; Metabolic Syndrome; Atherosclerosis; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After overnight fasting and supine rest for at least 10 minutes, blood was withdrawn from the antecubital vein. Serum was divided into aliquots and stored at -80°C.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The prevalence of metabolic syndrome in patients suffering from non valvular atrial fibrillation is derived from studies regarding recurrences of atrial fibrillation after catheter ablation. Prospective studies in european countries are lacking. Furthermore, the impact of metabolic syndrome on cardiovascular events in patients with non valvular atrial fibrillation is still unknown.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia that is associated with a high risk of cardiovascular events and increased morbidity and mortality. Cardiovascular events are prevalently localized in the cerebral circulation in which AF is responsible for ischemic stroke. Clinical characteristics of ischemic stroke from AF are almost severe and thromboembolism is considered the most important cause. Thus, ischemic stroke is deemed to origin from thrombus formation generated in the left atrium with ensuing embolism in the cerebral circulation.

Patients with AF are typically associated with different risk factors of atherothrombosis including, overall, hypertension which may be detected in about 70-80% of the population; other risk factors are diabetes and dyslipidemia. This accounts for instrumental evidence of systemic atherosclerosis associated to AF. Thus, signs of atherosclerosis have been detected in the thoracic aorta, as represented by aortic plaque assessed by trans-esophageal echocardiography; patients with complex aortic plaque had fourfold increased rate of stroke compared to plaque-free patients.

Metabolic syndrome (MetS) is a constellation of atherosclerotic risk factors including, according to the modified National Cholesterol Education Program Adult Treatment Panel III (NCEP-ATPIII), hypertension, low HDL, impaired glycaemic control, hypertriglyceridemia and central obesity as assessed by waist circumference; the presence of MetS is associated with an increased risk of developing cardiac and cerebral ischemic events.

An higher risk to develop atrial fibrillation (AF) has been well recognized in patients with MetS. In a prospective, community-based, observational cohort study with annual health check-up 28449 subjects without AF the age-adjusted rates of AF were higher in subjects with compared to those without metabolic syndrome during a mean follow-up of 4.5 years.

Few studies reported on the prevalence of MetS in AF population are still lacking. Some data can be inferred from studies regarding recurrence of AF after catheter ablation reporting a prevalence ranging from 18.8% to 49.4% . The only population study so far published included 741 chinese patients and reported a prevalence of the MetS in AF of 46.3%. Taking into account the thresholds of waist circumference recommended by international societies for different ethnic groups, it is unclear if such prevalence can be extrapolated to population of western countries.

Furthermore the impact of MetS on the incidence of cardiovascular events in patients with non valvular AF (NVAF) taking oral anticoagulant therapy (OAT) has never been investigated.

Therefore, our aim was to investigate the prevalence of MetS in a population of NVAF patients under oral coagulation treatment and its impact on cardiovascular events during a prospective study.

The study has been modified and approved by local ethical board of Sapienza University of Rome to include patients treated with non-vitamin K oral anticoagulants (dabigatran, apixaban, edoxaban, rivaroxaban) on April 11, 2014 (Prot. 417/14).

ELIGIBILITY:
Inclusion Criteria:

* non valvular atrial fibrillation
* age >18 years
* any antithrombotic treatment

Exclusion Criteria:

* prosthetic heart valves, or the presence of any severe valvulopathies, severe cognitive impairment, chronic infectious (HIV, hepatitis C, HBV) or autoimmune systemic disease. Furthermore, subjects were excluded from the study if they had active neoplastic diseases or liver insufficiency (eg, cirrhosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective single-center study including consecutive patients with NVAF referring to our center for monitoring and management of antithrombotic therapies of the Department of Internal Medicine and Medical Specialties of Sapienza-University of Rome from November 2007.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2007-11; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of metabolic syndrome in anticoagulated nonvalvular atrial fibrillation patients | At baseline
  To assess the prevalence of metabolic syndrome in a population of patients suffering from nonvalvular atrial fibrillation receiving oral anticoagulants. The relationship between metabolic syndrome and vascular events will be described. Vascular events included a composite outcome of fatal and non fatal acute myocardial infarction, acute fatal and non fatal ischemic stroke, cardiac revascularization (stent/cabg), cardiovascular death.

SECONDARY OUTCOMES:
Progression of atherosclerosis in non valvular atrial fibrillation patients receiving oral anticoagulant therapy. | One year
  To assess the progression of atherosclerosis in nonvalvular atrial fibrillation patients defined by some surrogate markers. In particular ankle brachial index, intima media thickness, flow mediated dilation and transthoracic echocardiogram will be performed to all enrolled patients.
Analysis of oxidative stress markers in atrial fibrillation | At baseline
  Oxidative stress markers such as plasmatic and urinary isoprostanes, thromboxane, platelet recruitment, reactive species of oxygen, nadph oxidase(nox2)will be measured. Differences of these markers among patients experiencing or not a vascular outcome will be described
Changing in glomerular filtration rate of anticoagulated patients with non valvular atrial fibrillation | One year
  To assess changes in renal function after one year of follow up in patients with non valvular atrial fibrillation receiving oral anticoagulants
Determinants of Time in Therapeutic Range | Patients will be followed for an expected mean time of 25 months
  To assess the determinants of time in therapeutic range (TTR) in patients receiving oral anticoagulants
Use of digoxin in atrial fibrillation | At baseline
  Use of digoxin will be assessed at baseline. The relationship with vascular outcomes will be described
Echocardiographic characteristics in patients with paroxysmal or persistent/permanent atrial fibrillation | At baseline
  Transthoracic echocardiography will be performed at baseline. Morphologic and functional measures will be registered. The relationship with vascular outcome will be described

OTHER OUTCOMES:
Mediterranean diet adherence in non valvular atrial fibrillation | At baseline
  To assess the adherence to the mediterranean diet in patients receiving oral anticoagulants

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, Prof, Study Director — Sapienza Università di Roma
Locations (1):
- Umberto I Policlinico di Roma, Sapienza Università di Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pignatelli P, Pastori D, Farcomeni A, Nocella C, Bartimoccia S, Vicario T, Bucci T, Carnevale R, Violi F. Mediterranean diet reduces thromboxane A2 production in atrial fibrillation patients. Clin Nutr. 2015 Oct;34(5):899-903. doi: 10.1016/j.clnu.2014.09.011. Epub 2014 Sep 28. PMID 25288566
- [Result] Pignatelli P, Pastori D, Carnevale R, Farcomeni A, Cangemi R, Nocella C, Bartimoccia S, Vicario T, Saliola M, Lip GY, Violi F. Serum NOX2 and urinary isoprostanes predict vascular events in patients with atrial fibrillation. Thromb Haemost. 2015 Mar;113(3):617-24. doi: 10.1160/TH14-07-0571. Epub 2014 Nov 13. PMID 25392853
- [Result] Pastori D, Pignatelli P, Angelico F, Farcomeni A, Del Ben M, Vicario T, Bucci T, Raparelli V, Cangemi R, Tanzilli G, Lip GYH, Violi F. Incidence of myocardial infarction and vascular death in elderly patients with atrial fibrillation taking anticoagulants: relation to atherosclerotic risk factors. Chest. 2015 Jun;147(6):1644-1650. doi: 10.1378/chest.14-2414. PMID 25429521
- [Result] Pastori D, Farcomeni A, Bucci T, Cangemi R, Ciacci P, Vicario T, Violi F, Pignatelli P. Digoxin treatment is associated with increased total and cardiovascular mortality in anticoagulated patients with atrial fibrillation. Int J Cardiol. 2015 Feb 1;180:1-5. doi: 10.1016/j.ijcard.2014.11.112. Epub 2014 Nov 18. PMID 25460369
- [Result] Pastori D, Carnevale R, Bartimoccia S, Nocella C, Tanzilli G, Cangemi R, Vicario T, Catena M, Violi F, Pignatelli P. Does Mediterranean Diet Reduce Cardiovascular Events and Oxidative Stress in Atrial Fibrillation? Antioxid Redox Signal. 2015 Sep 10;23(8):682-7. doi: 10.1089/ars.2015.6326. Epub 2015 Apr 28. PMID 25825798
- [Result] Pignatelli P, Pastori D, Vicario T, Bucci T, Del Ben M, Russo R, Tanzilli A, Nardoni ML, Bartimoccia S, Nocella C, Ferro D, Saliola M, Cangemi R, Lip GY, Violi F. Relationship between Mediterranean diet and time in therapeutic range in atrial fibrillation patients taking vitamin K antagonists. Europace. 2015 Aug;17(8):1223-8. doi: 10.1093/europace/euv127. Epub 2015 May 19. PMID 25995397
- [Result] Pastori D, Pignatelli P, Saliola M, Carnevale R, Vicario T, Del Ben M, Cangemi R, Barilla F, Lip GY, Violi F. Inadequate anticoagulation by Vitamin K Antagonists is associated with Major Adverse Cardiovascular Events in patients with atrial fibrillation. Int J Cardiol. 2015 Dec 15;201:513-6. doi: 10.1016/j.ijcard.2015.08.054. Epub 2015 Aug 5. PMID 26318513
- [Result] Pastori D, Pignatelli P, Farcomeni A, Cangemi R, Hiatt WR, Bartimoccia S, Nocella C, Vicario T, Bucci T, Carnevale R, Lip GY, Violi F. Urinary 11-dehydro-thromboxane B2 is associated with cardiovascular events and mortality in patients with atrial fibrillation. Am Heart J. 2015 Sep;170(3):490-7.e1. doi: 10.1016/j.ahj.2015.05.011. Epub 2015 May 22. PMID 26385032
- [Result] Pastori D, Farcomeni A, Poli D, Antonucci E, Angelico F, Del Ben M, Cangemi R, Tanzilli G, Lip GY, Pignatelli P, Violi F. Cardiovascular risk stratification in patients with non-valvular atrial fibrillation: the 2MACE score. Intern Emerg Med. 2016 Mar;11(2):199-204. doi: 10.1007/s11739-015-1326-1. Epub 2015 Oct 15. PMID 26471883
- [Result] Pastori D, Pignatelli P, Perticone F, Sciacqua A, Carnevale R, Farcomeni A, Basili S, Corazza GR, Davi G, Lip GYH, Violi F; ARAPACIS (Atrial Fibrillation Registry for Ankle-Brachial Index Prevalence Assessment-Collaborative Italian Study) study group. Aspirin and renal insufficiency progression in patients with atrial fibrillation and chronic kidney disease. Int J Cardiol. 2016 Nov 15;223:619-624. doi: 10.1016/j.ijcard.2016.08.224. Epub 2016 Aug 14. PMID 27565838
- [Result] Pastori D, Pignatelli P, Farcomeni A, Menichelli D, Nocella C, Carnevale R, Violi F. Aging-Related Decline of Glutathione Peroxidase 3 and Risk of Cardiovascular Events in Patients With Atrial Fibrillation. J Am Heart Assoc. 2016 Sep 8;5(9):e003682. doi: 10.1161/JAHA.116.003682. PMID 27609361
- [Result] Pastori D, Pignatelli P, Farcomeni A, Nocella C, Bartimoccia S, Carnevale R, Violi F. Age-related increase of thromboxane B2 and risk of cardiovascular disease in atrial fibrillation. Oncotarget. 2016 Jun 28;7(26):39143-39147. doi: 10.18632/oncotarget.9826. PMID 27270651
- [Result] Pastori D, Carnevale R, Menichelli D, Nocella C, Bartimoccia S, Novo M, Leo I, Violi F, Pignatelli P. Is There an Interplay Between Adherence to Mediterranean Diet, Antioxidant Status, and Vascular Disease in Atrial Fibrillation Patients? Antioxid Redox Signal. 2016 Nov 10;25(14):751-755. doi: 10.1089/ars.2016.6839. Epub 2016 Sep 30. PMID 27577528
- [Result] Pastori D, Carnevale R, Nocella C, Novo M, Santulli M, Cammisotto V, Menichelli D, Pignatelli P, Violi F. Gut-Derived Serum Lipopolysaccharide is Associated With Enhanced Risk of Major Adverse Cardiovascular Events in Atrial Fibrillation: Effect of Adherence to Mediterranean Diet. J Am Heart Assoc. 2017 Jun 5;6(6):e005784. doi: 10.1161/JAHA.117.005784. PMID 28584074
- [Result] Carnevale R, Pignatelli P, Frati G, Nocella C, Stanzione R, Pastori D, Marchitti S, Valenti V, Santulli M, Barbato E, Strisciuglio T, Schirone L, Vecchione C, Violi F, Volpe M, Rubattu S, Sciarretta S. C2238 ANP gene variant promotes increased platelet aggregation through the activation of Nox2 and the reduction of cAMP. Sci Rep. 2017 Jun 19;7(1):3797. doi: 10.1038/s41598-017-03679-9. PMID 28630469
- [Result] Pastori D, Nocella C, Farcomeni A, Bartimoccia S, Santulli M, Vasaturo F, Carnevale R, Menichelli D, Violi F, Pignatelli P; ATHERO-AF Study Group. Relationship of PCSK9 and Urinary Thromboxane Excretion to Cardiovascular Events in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2017 Sep 19;70(12):1455-1462. doi: 10.1016/j.jacc.2017.07.743. PMID 28911508
- [Result] Pastori D, Pignatelli P, Sciacqua A, Perticone M, Violi F, Lip GYH. Relationship of peripheral and coronary artery disease to cardiovascular events in patients with atrial fibrillation. Int J Cardiol. 2018 Mar 15;255:69-73. doi: 10.1016/j.ijcard.2017.12.076. Epub 2017 Dec 24. PMID 29290420
- [Derived] Baratta F, Bartimoccia S, Pastori D, Cocomello N, Cammisotto V, Castellani V, Nocella C, Forte M, Picchio V, Carnevale R, Desideri G, Pignatelli P, Violi F. Neutrophil cathepsin G and risk of cardiovascular events in patients with diabetes mellitus. Cardiovasc Diabetol. 2025 Nov 26;24(1):448. doi: 10.1186/s12933-025-03005-y. PMID 41299502
- [Derived] Pastori D, Menichelli D, Lip GYH, Sciacqua A, Violi F, Pignatelli P; ATHERO-AF study groupdagger. Family History of Atrial Fibrillation and Risk of Cardiovascular Events: A Multicenter Prospective Cohort Study. Circ Arrhythm Electrophysiol. 2020 Sep;13(9):e008477. doi: 10.1161/CIRCEP.120.008477. Epub 2020 Jul 27. PMID 32718257
- [Derived] Pastori D, Pignatelli P, Menichelli D, Violi F, Lip GYH. Integrated Care Management of Patients With Atrial Fibrillation and Risk of Cardiovascular Events: The ABC (Atrial fibrillation Better Care) Pathway in the ATHERO-AF Study Cohort. Mayo Clin Proc. 2019 Jul;94(7):1261-1267. doi: 10.1016/j.mayocp.2018.10.022. Epub 2018 Dec 11. PMID 30551910
- [Derived] Pastori D, Carnevale R, Cangemi R, Saliola M, Nocella C, Bartimoccia S, Vicario T, Farcomeni A, Violi F, Pignatelli P. Vitamin E serum levels and bleeding risk in patients receiving oral anticoagulant therapy: a retrospective cohort study. J Am Heart Assoc. 2013 Oct 28;2(6):e000364. doi: 10.1161/JAHA.113.000364. PMID 24166490